CLINICAL TRIAL: NCT02768688
Title: Glymphatic Clearance During Anesthesia and Sleep: A Diffusion Tensor Imaging (DTI) Study in Humans
Brief Title: MRI of Glymphatic Clearance During Anesthetic Sedation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 819962
Record Dates: First submitted 2016-04-05; First posted 2016-05-11 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Glymphatic Flow
Keywords: Human Brain; Magnetic Resonance Imaging (MRI); Dexmedetomidine; Cerebral blood flow
MeSH Terms: interventions — Functional Status; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brain connectivity and physiology (Experimental): Dexmedetomidine anesthesia on glymphatic flow in human subjects as visualized by diffusion tensor MRI.
  Interventions: Other: Brain connectivity and physiology; Drug: Dexmedetomidine

INTERVENTIONS:
Other: Brain connectivity and physiology — MRI to measure glymphactic flow during simulated natural sleep and again on return to wakefulness.
Drug: Dexmedetomidine — Administering of 0.5-1.0 mcg/kg/hr of dexmedetomidine to ensure subject's loss of consciousness.

SUMMARY:
This study is to assess the effect of dexmedetomidine anesthesia on glymphatic flow in 5 healthy human subjects as visualized by diffusion tensor MRI. The study is designed to measure clinically established, safe imaging of DTI and cerebral blood flow at baseline, during a continuous intravenous infusion of dexmedetomidine at doses designed to produce anesthesia-induced unconsciousness to simulate natural sleep, and again on return to wakefulness.

DETAILED DESCRIPTION:
Objective:

The purpose of this study is to assess the effect of dexmedetomidine anesthesia on glymphatic flow in human subjects as visualized by diffusion tensor MRI.

Study Design:

This study will take place at the University of Pennsylvania. Investigators plan to enroll approximately 30 healthy volunteers to generate pilot data for a larger grant submission.

Characteristics of the Study Population:

Subjects will be healthy males or females aged 20 to 40 years of age who will be recruited to participate in an MRI scan designed to measure clinically established, safe imaging of diffusion tensor imaging and cerebral blood flow at baseline, during a continuous intravenous infusion of dexmedetomidine at doses designed to produce anesthesia-induced unconsciousness to simulate natural sleep, and again on return to wakefulness. They must be able to pass the standard MRI safety assessment (e.g., no metallic metal clips or implants or any other contraindications to undergoing an MRI).

Design:

Upon successful completion of screening questionnaire, urine drug, and urine pregnancy subjects will be scheduled for an MRI. On the day of the study subjects will receive an intravenous catheter (IV) for study drug and fluids. Set one of MRI scans will be done with no dexmedetomidine. Set two of scans will be done when subject is anesthetized with dexmedetomidine with the goal depth of sedation will be moderate sedation. Set three of scans will be done when dexmedetomidine is stopped and wakefulness is achieved.

ELIGIBILITY:
Inclusion Criteria:

1. Person aged 20-40 years old,
2. American Society of Anesthesiologists Physical Status I or II (i.e., healthy),
3. Body mass index ≤ 30 kg/m2,
4. Easily visualized uvula,
5. Not a current tobacco user
6. No history of alcohol abuse/must abstain from alcohol use 24 hours prior to and 24 hours after participation.
7. Ability to sign informed consent.
8. Able to pass standard MRI safety screening
9. Must have a responsible adult available to transport subject home safely after end of experiment.

Exclusion Criteria:

1. Healthy male or females less than 20 years of age or older than 40 years of age
2. Any physical signs suggestive of difficult airway (mouth opening 3cm, short distance between the chin and neck, poor mandibular subluxation, thick neck),
3. History of obstructive sleep apnea,
4. History of asthma
5. Neuropsychiatric disorders,
6. History of, or current use of psychotropic medications,
7. Current tobacco use or history of smoking in past month
8. Alcohol use exceeding 2 drinks/day
9. History of hypertension or current medication for blood pressure control,
10. Cardiovascular disease or arrhythmias,
11. Positive urine toxicology screen,
12. History of gastroesophageal reflux disease,
13. Pregnancy,
14. Sleep disorders,
15. History of postoperative nausea/vomiting or motion sickness,
16. Inability to sign informed consent
17. Contraindications for safely participating in MRI imaging study,
18. Does not have a responsible adult available to provide transport from HUP MRI area to home.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2014-07; Primary Completion 2017-02-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Glymphatic clearance from the human brain | 2 hours
  Assessment of the effect of dexmedetomidine anesthesia on glymphatic flow in subjects as visualized by diffusion tensor MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Max B Kelz, MD, Principal Investigator — Physician
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No